CLINICAL TRIAL: NCT00990054
Title: A Phase I, Dose Escalation Study of Plerixafor in Combination With Cytarabine and Daunorubicin in Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Study of Plerixafor Combined With Cytarabine and Daunorubicin in Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOZ04808
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Cytarabine,; Daunorubicin,; De Novo,; Acute Myeloid Leukemia,; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- plerixafor (Experimental)
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — 240 mcg/kg/dose and proceeding to escalating dose levels for determination of the single-dose maximum tolerated dose (MTD) provided that there are no unacceptable dose limiting toxicities
  Other Names: AMD3100; Mozobil

SUMMARY:
The purpose of this research study is to determine if plerixafor can make cells more sensitive to killing by cytarabine and daunorubicin, an anti-cancer drug regimen referred to as "7+3" that is commonly used in treating acute myeloid leukemia (AML). In this study, plerixafor is used with treatments cytarabine and daunorubicin and with and without granulocyte-colony stimulating factor (GCSF). Subjects will be monitored to see how well they tolerate the use of these drugs together and how well they work to treat the leukemia.

The purpose of the study is to determine the maximum tolerated dose (MTD) per plerixafor dosing schedule (once daily [QD] or twice daily [BID]), and/or recommended phase 2 dose (RP2D), by assessing safety and tolerability of plerixafor (Mozobil®) when used in combination with cytarabine and daunorubicin, and with and without granulocyte-colony stimulating factor (G-CSF)

ELIGIBILITY:
Inclusion Criteria:

* Provide signed, dated informed consent prior to any protocol-specific procedures.
* Have a diagnosis of newly diagnosed AML, defined as >20% myeloblasts on the marrow aspirate or peripheral blood differential, with or without extramedullary involvement, with confirmatory immunophenotyping or immunocytochemistry (e.g., myeloperoxidase), documented within 14 days of enrollment.
* Have Eastern Cooperative Oncology Group (ECOG) performance status (Appendix A) score of 0, 1, or 2.
* Toxicities from all prior treatments have resolved to baseline or δ Grade 1 prior to first dose of study drugs.
* Are surgically or biologically sterile or willing to practice acceptable birth control, as follows: Females of child bearing potential must agree to abstain from sexual activity or to use a medically approved contraceptive measure/regimen during and for 3 months after the treatment period. Women of child bearing potential must have a negative serum pregnancy test at the time of enrollment. Acceptable methods of birth control include oral contraceptive, intrauterine device (IUD), transdermal/implanted or injected contraceptives and abstinence.
* Males must agree to abstain from sexual activity or agree to utilize a medially-approved contraception method during and for 3 months after the treatment period.
* Have adequate renal and hepatic function, as indicated by the following laboratory values: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) δ2.5 - upper limit of normal (ULN); Estimated creatinine clearance (CrCl) of > 50mL/min, as calculated by the Cockcroft-Gault equation (Appendix F); total bilirubin ≤1.5-ULN (except in patients with Gilbert Syndrome, in whom direct bilirubin must be ≤1.5-ULN), International Normalized Ratio (INR) ≤1.5 after discontinuation of anticoagulants.
* Have adequate cardiac function, as measured by left ventricular ejection fraction (LVEF) ≥40% on echocardiography or multigated acquisition (MUGA) scan or similar radionuclide angiographic scan.
* Be able to comply with study procedures and follow-up examinations.

Exclusion Criteria:

* Have received previous systemic treatment for leukemia or antecedent hematologic disorder (AHD), other than hydroxyurea or hematopoietic growth factors. Treatment with hydroxyurea within 2 weeks of screening is allowed but must be discontinued at least 24 hours prior to the first dose of study drugs.
* Have received prior treatment with plerixafor, cytarabine, or any anthracycline.
* Have a diagnosis of acute promyelocytic leukemia (APL), French-American-British (FAB) classification M3 or World Health Organization (WHO) classification of APL with t(15;17)(q(22;q12), or Bcr-Abl positive leukemia.
* For patients < 50 years of age, have cytogenetics associated with good prognosis [(t(8;21)q(22;22), t(15;17),inv(16)(p13;q22)]. (Testing for these mutations must be performed on blood or Bone Marrow prior to study registration.
* Have had a hematopoietic stem cell transplant (HSCT).
* Have an absolute blast count of the following at the time of first dose of chemotherapy, despite cytoreduction with hydroxyurea or leukapheresis:

  1. >50 x 10^9/L for patients not enrolled in a G-CSF-containing cohort
  2. >25 x 10^9/L for patients enrolled in a G-CSF-containing cohort
* Have central nervous system (CNS) leukemia (Only patients with suspected CNS leukemia must undergo lumbar puncture.)
* Have any of the following within the last 12 months: unstable supraventricular arrhythmia (e.g., hemodynamic instability) or has a pacemaker; Any ventricular arrhythmia, other than occasional premature ventricular contractions; Congestive heart failure (controlled or uncontrolled); Myocardial infarction, ischemia, stable coronary artery disease, or angina; Uncontrolled hypertension; Syncope with either a known cardiovascular or an unknown etiology.
* Have a pre-existing disorder predisposing the patient to serious or life-threatening infection (e.g., cystic fibrosis, congenital or acquired immunodeficiency, bleeding disorder, or cytopenias).
* Have the need for anticoagulant therapy.
* Have a significant medical or psychiatric disorder that would interfere with consent, study participation, or follow-up.
* Have an active acute or chronic systemic fungal, bacterial, viral, or other infection (i.e., exhibiting ongoing signs/symptoms related to the infection [except isolated fever] and without improvement, despite appropriate antibiotics or other treatment).
* Have severe concurrent diseases (e.g., a history of serious organ dysfunction or disease) that may place the patient at undue risk to undergo induction therapy per protocol, or obscure assessments of drug safety.
* Have a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent, with the following exceptions:

  1. Patients with treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, if definitive treatment for the condition has been completed; or
  2. Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values after treatment with curative intent.
* Have known human immunodeficiency virus (HIV) positivity or evidence of active viral hepatitis.
* Are pregnant or breastfeeding.
* Are known to have an allergy to any component of the study drug regimen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of plerixafor when used in combination with cytarabine and daunorubicin and with and without GCSF | 28 days from first dose and up to 42 days following last dose

SECONDARY OUTCOMES:
Anti-leukemia activity of plerixafor when used with cytarabine and daunorubicin | Beginning at Day 14 and then until complete remission (CR), complete remission with incomplete count recovery (CRi), or treatment failure (TF)
Maximal plasma concentration (Cmax) of plerixafor when used with cytarabine and daunorubicin | Cycle 1 (1 week)
Time to maximal plasma concentration (Tmax) of Plerixafor when used with cytarabine and daunorubicin | Cycle 1 (1 week)
Area under the concentration-time curve from time zero to the last observed concentration (AUC 0-last) of plerixafor when used with cytarabine and daunorubicin | Cycle 1 (1 week)
Area under the concentration-time curve over the dosing interval (τ) (AUC 0-τ) of plerixafor when used with cytarabine and daunorubicin | Cycle 1 (1 week)
Area under the concentration-time curve from time zero to infinity (AUC 0-∞ ) of plerixafor when used with cytarabine and daunorubicin | Cycle 1 (1 week)
Half-life (T½) of plerixafor when used with cytarabine and daunorubicin | Cycle 1 (1 week)
Volume of distribution (Vz/F for SC administration; Vz for IV administration); in the case of multiexponential disposition, volume of distribution at steady-state (Vss) will be calculated of plerixafor when used with cytarabine and daunorubicin | Cycle 1 (1 week)
Obtain preliminary data on safety , tolerability, PK, leukemia cell mobilization and anti-leukemia activity of plerixafor when used in conjunction with G-CSF, cytarabine and daunorubicin. | Cycle 1 (1 week) and then until complete remission (CR), complete remission with incomplete count recovery (CRi), or treatment failure (TF)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (8):
  - Duarte, California
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Rochester, New York
  - Cleveland, Ohio
  - Houston, Texas
  - Seattle, Washington